CLINICAL TRIAL: NCT02122146
Title: A Phase 1, Dose Escalation Study Of Pf-06664178 In Patients With Locally Advanced Or Metastatic Solid Tumors
Brief Title: A Study Of PF-06664178 In Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was prematurely discontinued due to a business-related decision on 09-FEB-2016. The decision to terminate the trial was based on the overall results.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: B7401001; 2015-002704-84 (EudraCT Number)
Record Dates: First submitted 2014-04-17; First posted 2014-04-24 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2017-08

CONDITIONS: Neoplasms
Keywords: ADC; PF-06664178; solid tumors; tumors; neoplasm metastasis; NSCLC; non small cell lung cancer; OVCA; ovarian cancer; Phase 1; breast cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-06664178 (Experimental): Experimental
  Interventions: Drug: PF-06664178

INTERVENTIONS:
Drug: PF-06664178 — Part 1 - PF-06664178 will be administered intravenously every 21 days in cohorts of 2 or more patients starting at a dose of 0.15 mg/kg. Increases in dose will continue until MTD is determined.
Drug: PF-06664178 — Part 2 - patients with select tumor types (Non Small Cell Lung Cancer ovarian cancer, and breast cancer ) will be treated at the MTD selected in Part 1.

SUMMARY:
To assess the safety and tolerability at increasing dose levels of PF-06664178 in patients with advanced solid tumors in order to determine the maximum tolerated dose and select the recommended Phase 2 dose.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of solid tumor that is advanced/metastatic and resistant to standard therapy or for whom no standard therapy is available
* Performance Status of 0 or 1
* Adequate bone marrow, kidney and liver function
* Part 2 includes target expressing NSCLC, ovarian or breast cancer patients

Exclusion Criteria:

* Brain metastases requiring steroids
* Major surgery, radiation therapy, or systemic anti-cancer therapy within 4 weeks of study treatment start (6 weeks for mitomycin C or nitrosoureas)
* Active and clinically significant bacterial, fungal, or viral infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (10):
  - Keck Hospital of USC, Los Angeles, California
  - LAC&USC Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center / Investigational Drug Services, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Colorado Denver CTO (CTRC), Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Swedish Medical Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7401001&StudyName=A%20Study%20Of%20PF-06664178%20In%20Patients%20With%20Advanced%20Solid%20Tumors

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 38 patients were screened, among which 31 were assigned to study treatment.
Groups:
- PF-06664178 0.15 mg/kg: Participants were enrolled in cohorts of 2-4 to receive PF-06664178 in an open-label, unblinded manner and treated with PF-06664178 in 7 sequential dose levels between 0.15 and 4.8 mg/kg. PF-06664178 0.15 mg/kg was administered on Day 1 of each 21-day cycle per the dose administration instructions (DAI) as an intravenous (IV) infusion over 60 minutes ±5 minutes on an outpatient basis.
- PF-06664178 0.30 mg/kg: Participants were enrolled in cohorts of 2-4 to receive PF-06664178 in an open-label, unblinded manner and treated with PF-06664178 in 7 sequential dose levels between 0.15 and 4.8 mg/kg. PF-06664178 0.30 mg/kg was administered on Day 1 of each 21-day cycle per the DAI as an IV infusion over 60 minutes ±5 minutes on an outpatient basis.
- PF-06664178 0.60 mg/kg: Participants were enrolled in cohorts of 2-4 to receive PF-06664178 in an open-label, unblinded manner and treated with PF-06664178 in 7 sequential dose levels between 0.15 and 4.8 mg/kg. PF-06664178 0.60 mg/kg was administered on Day 1 of each 21-day cycle per the DAI as an IV infusion over 60 minutes ±5 minutes on an outpatient basis.
- PF-06664178 1.20 mg/kg: Participants were enrolled in cohorts of 2-4 to receive PF-06664178 in an open-label, unblinded manner and treated with PF-06664178 in 7 sequential dose levels between 0.15 and 4.8 mg/kg. PF-06664178 1.20 mg/kg was administered on Day 1 of each 21-day cycle per the DAI as an IV infusion over 60 minutes ±5 minutes on an outpatient basis.
- PF-06664178 2.40 mg/kg: Participants were enrolled in cohorts of 2-4 to receive PF-06664178 in an open-label, unblinded manner and treated with PF-06664178 in 7 sequential dose levels between 0.15 and 4.8 mg/kg. PF-06664178 2.40 mg/kg was administered on Day 1 of each 21-day cycle per the DAI as an IV infusion over 60 minutes ±5 minutes on an outpatient basis.
- PF-06664178 3.60 mg/kg: Participants were enrolled in cohorts of 2-4 to receive PF-06664178 in an open-label, unblinded manner and treated with PF-06664178 in 7 sequential dose levels between 0.15 and 4.8 mg/kg. PF-06664178 3.60 mg/kg was administered on Day 1 of each 21-day cycle per the DAI as an IV infusion over 60 minutes ±5 minutes on an outpatient basis.
- PF-06664178 4.20 mg/kg: Participants were enrolled in cohorts of 2-4 to receive PF-06664178 in an open-label, unblinded manner and treated with PF-06664178 in 7 sequential dose levels between 0.15 and 4.8 mg/kg. PF-06664178 4.20 mg/kg was administered on Day 1 of each 21-day cycle per the DAI as an IV infusion over 60 minutes ±5 minutes on an outpatient basis.
- PF-06664178 4.80 mg/kg: Participants were enrolled in cohorts of 2-4 to receive PF-06664178 in an open-label, unblinded manner and treated with PF-06664178 in 7 sequential dose levels between 0.15 and 4.8 mg/kg. PF-06664178 4.80 mg/kg was administered on Day 1 of each 21-day cycle per the DAI as an IV infusion over 60 minutes ±5 minutes on an outpatient basis.
Period: Part 1: Dose Escalation
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Started | 2 | 2 | 4 | 4 | 4 | 6 | 1 | 8
Completed | 1 | 1 | 2 | 3 | 3 | 5 | 0 | 6
Not Completed | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 2
Not completed — Death | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Period: Part 2: Maximum Tolerated Dose
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Started | 0 (No participant enrolled due to study termination) | 0 (No participant enrolled due to study termination) | 0 (No participant enrolled due to study termination) | 0 (No participant enrolled due to study termination) | 0 (No participant enrolled due to study termination) | 0 (No participant enrolled due to study termination) | 0 (No participant enrolled due to study termination) | 0 (No participant enrolled due to study termination)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3: Expansion
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Started | 0 (No participant enrolled due to study termination) | 0 (No participant enrolled due to study termination) | 0 (No participant enrolled due to study termination) | 0 (No participant enrolled due to study termination) | 0 (No participant enrolled due to study termination) | 0 (No participant enrolled due to study termination) | 0 (No participant enrolled due to study termination) | 0 (No participant enrolled due to study termination)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg | Total
Number analyzed (Participants) | 2 | 2 | 4 | 4 | 4 | 6 | 1 | 8 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (7.1) | 75 (11.3) | 61 (17.9) | 52.8 (20) | 46 (11) | 53.7 (11.8) | 63 (0) | 61.1 (6.6) | 57.1 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 2 | 1 | 5 | 1 | 6 | 18
  Male | 1 | 2 | 2 | 2 | 3 | 1 | 0 | 2 | 13

OUTCOME MEASURES:

1. Primary Outcome: First Cycle Dose Limiting Toxicities (DLTs) In Order to Determine the Maximum Tolerated Dose(MTD)
Description: Number of participants that experienced dose limiting toxicities(DLTs) at given dose level.
Time Frame: Day 1 up to Day 21
Population: All enrolled participants who started treatment. One of participants that experienced DLTs in PF-06664178 4.80mg/kg group was a late DLT that occurred at the beginning of Cycle 2 and was classified as a late DLT.
Measure: Number; unit: participants
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 2 | 2 | 4 | 4 | 4 | 6 | 1 | 8
participants
  Yes | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 4
  No | 2 | 2 | 4 | 4 | 4 | 4 | 0 | 4

2. Primary Outcome: Number of Patients With All-Causality Treatment-Emergent Adverse Events(TEAEs) [Part 2 & 3]
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation subject administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. TEAEs were those AEs with initial onset or increasing in severity after the first dose of study drug.
Time Frame: Day 1 up to Day 21
Population: No participant was analyzed due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Laboratory Abnormalities [Part 2 & 3]
Description: Number of participants with a laboratory abnormality meeting specified criteria. The laboratory test included: hematology( hemoglobin, platelets, white blood cell count, absolute neutrophils, absolute lymphocytes, absolute monocytes, absolute eosinophils, absolute basophils), chemistry (alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, sodium, potassium, magnesium, chloride, total calcium, total bilirubin, blood urea nitrogen or urea, creatinine, uric acid, glucose, albumin, phosphorous or phosphate), coagulation (prothrombin time or International normalized ratio, partial thromboplastin time), Urinalysis (urine protein, urine blood) and pregnancy test.
Time Frame: On Day1, Day4, Day8, Day15 of the first cycle; on Day1, Day8, Day15 of the second cycle; on Day 1 of the subsequent cycles; end of treatment visit(no longer than 1 week after the patient has been discontinued)
Population: No participant was analyzed due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With All-Causality Treatment-Emergent Adverse Events (TEAEs ) [Part 1]
Description: as for outcome 2
Time Frame: From screening up to 28 days after the last treatment administration in each cycle, and follow-up visits(At least 28 days and no more than 35 days after discontinuation of treatment)
Population: All enrolled participants who started treatment
Measure: Number; unit: participants
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 2 | 2 | 4 | 4 | 4 | 6 | 1 | 8
participants | 2 | 2 | 4 | 4 | 4 | 6 | 1 | 8

5. Secondary Outcome: Number of Participants With Laboratory Abnormalities[Part 1]
Description: as for outcome 3
Time Frame: Screening; on Day1, Day4, Day8, Day15 of the first cycle; on Day1, Day8, Day15 of the second cycle; on Day 1 of the subsequent cycles; end of treatment visit(no longer than 1 week after the patient has been discontinued)
Population: All enrolled participants who started treatment.
Measure: Number; unit: participants
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 2 | 2 | 4 | 4 | 4 | 6 | 1 | 8
participants | 1 | 2 | 4 | 4 | 4 | 6 | 0 | 8

6. Secondary Outcome: Overall Incidence of Anti-PF-06664178-Antibodies[Part 1]
Description: Number of participants with the presence of anti-PF-06664178 antibodies
Time Frame: Day 1, 15, 21, and every 21 days thereafter up to 24 months, and end of treatment
Population: All enrolled participants who started treatment
Measure: Number; unit: participants
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 2 | 2 | 4 | 4 | 4 | 6 | 1 | 8
participants | 2 | 2 | 4 | 4 | 4 | 6 | 0 | 8

7. Secondary Outcome: Overall Incidence of Anti-PF-06664178-Antibodies [Part 2 & 3]
Description: Number of participants with the presence of anti-PF-06664178 antibodies
Time Frame: Day 1, 15, 21, and every 21 days thereafter up to 24 months, and end of treatment
Population: No participant was analyzed due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Overall Number of Participants With Objective Tumor Response[Part 1]
Description: Objective tumor response, was assessed using the Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1 by calculating the Overall Response Rate, and Prolonged Stable Disease. The criterion is defined as: Objective Progression(PD):20% increase in the sum of diameters of target measurable lesions above the smallest sum observed, with a minimum absolute increase of 5mm; Stable (SD): All target lesions must be assessed. Stable can follow PR only in the rare case that the sum increases by less than 20% from the nadir, but enough that a previously documented 30% decrease no longer holds; symptomatic deterioration(Sym):Participants with a global deterioration of health status requiring discontinuation of treatment without objective evidence of disease progression at that time; Indeterminate (In):Progression has not been determined and one, or more non-target sites were not assessed, or assessment methods were inconsistent with those used at baseline.
Time Frame: Baseline, every 6 weeks until disease progression or unacceptable toxicity up to 24 months
Population: Of all enrolled 31 patients who were treated, 1 participant from the 0.60mg/kg cohort and 1 participant from the 4.20mg/kg cohort did not have post-dose tumor evaluations for they were discontinued form study prior to having disease assessment .
Measure: Number; unit: participants
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 2 | 2 | 3 | 4 | 4 | 6 | 0 | 8
participants
  SD | 0 | 1 | 1 | 1 | 2 | 4 |  | 2
  PD | 2 | 1 | 2 | 3 | 2 | 1 |  | 3
  Sym | 0 | 0 | 0 | 0 | 0 | 1 |  | 0
  In | 0 | 0 | 0 | 0 | 0 | 0 |  | 3

9. Secondary Outcome: Overall Number of Participants With Objective Tumor Response [Part 2 & 3]
Description: Objective tumor response, as assessed using the Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1 by calculating the Overall Response Rate (ORR), and Prolonged Stable Disease (SD).No Progression Free Survival (PFS) was completed. The criterion is as follow: Objective Progression(PD), Stable (SD), symptomatic deterioration(Sym), and Indeterminate (In)
Time Frame: Baseline, every 6 weeks until disease progression or unacceptable toxicity up to 24 months
Population: No participant was analyzed due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for PF-06664178 [Part 1 ,2 & 3]
Description: Cmax of PF-06664178 was observed directly from data
Time Frame: 0, 1, 4, 24 hours post-dose on Day 1, and on Day 4, Day 8 and Day 15 of cycles 1 and 4; 0, 1hour post-dose on Cycle 2, 3 and every cycle after cycle 4, end of treatment
Population: Data were not collected during Part 1, and no participant was analyzed in Part 2 and 3 due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Total Antibody (PF-06479118) [Part 1 ,2 & 3]
Description: Cmax of total antibody PF-06479118 was observed directly from data
Time Frame: as for outcome 10
Population: Data were not collected during Part 1, and no participant was analyzed in Part 2 and 3 due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Unconjugated Payload (PF-06380101) [Part 1 ,2 & 3]
Description: Cmax of unconjugated payload PF-06380101 was observed directly from data
Time Frame: as for outcome 10
Population: Data were not collected during Part 1, and no participant was analyzed in Part 2 and 3 due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Area Under the Concentration-Time Curve Over the Dosing Interval(AUCtau) of PF-06664178 [Part 1 ,2 & 3]
Description: AUCtau refers to area under the concentration-time profile from time zero to the time tau, the dosing interval
Time Frame: as for outcome 10
Population: Data were not collected during Part 1, and no participant was analyzed in Part 2 and 3 due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Area Under the Concentration-Time Curve Over the Dosing Interval(AUCtau) of Total Antibody(PF-06479118) [Part 1 ,2 & 3]
Description: AUCtau refers to area under the concentration-time profile from time zero to the time tau, the dosing interval.
Time Frame: as for outcome 10
Population: Data were not collected during Part 1, and no participant was analyzed in Part 2 and 3 due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Area Under the Concentration-Time Curve Over the Dosing Interval(AUCtau) of Unconjugated Payload(PF-06380101) [Part 1 ,2 & 3]
Description: AUCtau refers to area under the concentration-time profile from time zero to the time tau, the dosing interval.
Time Frame: as for outcome 10
Population: Data were not collected during Part 1, and no participant was analyzed in Part 2 and 3 due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Systemic Clearance (CL) of PF-06664178 [Part 1 ,2 & 3]
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: as for outcome 10
Population: Data were not collected during Part 1, and no participant was analyzed in Part 2 and 3 due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Systemic Clearance (CL) of Total Antibody (PF-06479118) [Part 1 ,2 & 3]
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: as for outcome 10
Population: Data were not collected during Part 1, and no participant was analyzed in Part 2 and 3 due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Systemic Clearance (CL) of Unconjugated Payload (PF-06380101) [Part 1 ,2 & 3]
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: as for outcome 10
Population: Data were not collected during Part 1, and no participant was analyzed in Part 2 and 3 due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Volume of Distribution (Vss) of PF-06664178 [Part 1 ,2 & 3]
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.
Time Frame: as for outcome 10
Population: Data were not collected during Part 1, and no participant was analyzed in Part 2 and 3 due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Volume of Distribution (Vss) of Total Antibody (PF-06479118) [Part 1 ,2 & 3]
Description: as for outcome 19
Time Frame: as for outcome 10
Population: Data were not collected during Part 1, and no participant was analyzed in Part 2 and 3 due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Volume of Distribution (Vss) of Unconjugated Payload (PF-06380101) [Part 1 ,2 & 3]
Description: as for outcome 19
Time Frame: as for outcome 10
Population: Data were not collected during Part 1, and no participant was analyzed in Part 2 and 3 due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of PF-06664178 [Part 1 ,2 & 3]
Description: Terminal elimination half-life is the time measured for the plasma concentration to decrease by one half
Time Frame: as for outcome 10
Population: Data were not collected during Part 1, and no participant was analyzed in Part 2 and 3 due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of Total Antibody (PF-06479118)[Part 1 ,2 & 3]
Description: Terminal elimination half-life is the time measured for the plasma concentration to decrease by one half
Time Frame: as for outcome 10
Population: Data were not collected during Part 1, and no participant was analyzed in Part 2 and 3 due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of Unconjugated Payload (PF-06380101) [Part 1 ,2 & 3]
Description: Terminal elimination half-life is the time measured for the plasma concentration to decrease by one half
Time Frame: as for outcome 10
Population: Data were not collected during Part 1, and no participant was analyzed in Part 2 and 3 due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Trop-2 Expression Levels on Archived Tissue [Part 2 & 3]
Description: Number of participents meeting the following criterion for Trop-2 expression assessment : low expression, medium expression and high expression
Time Frame: Day 1
Population: No participant was analyzed due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Accumulation Ratio (Rac) of PF-06664178 [Part 1 ,2 & 3]
Description: Accumulation ratio refers to AUCtau for cycle 4/AUCtau for cycle 1, where AUCtau is defined as area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to the time tau, the dosing interval.
Time Frame: as for outcome 10
Population: Data were not collected during Part 1, and no participant was analyzed in Part 2 and 3 due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Accumulation Ratio (Rac) of Total Antibody (PF-06479118) [Part 1 ,2 & 3]
Description: as for outcome 26
Time Frame: as for outcome 10
Population: Data were not collected during Part 1, and no participant was analyzed in Part 2 and 3 due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: Accumulation Ratio (Rac) of Unconjugated Payload (PF-06380101) [Part 1 ,2 & 3]
Description: as for outcome 26
Time Frame: as for outcome 10
Population: Data were not collected during Part 1, and no participant was analyzed in Part 2 and 3 due to study termination
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From screening up to 28 days after the last treatment administration in each cycle, and follow-up visits(at least 28 days and no more than 35 days after discontinuation of treatment)
Groups:
- Total: Treatment Group Description TBD
Arm/Group | PF-06664178 0.15 mg/kg | PF-06664178 0.30 mg/kg | PF-06664178 0.60 mg/kg | PF-06664178 1.20 mg/kg | PF-06664178 2.40 mg/kg | PF-06664178 3.60 mg/kg | PF-06664178 4.20 mg/kg | PF-06664178 4.80 mg/kg | Total
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/2 | 2/4 | 0/4 | 1/4 | 3/6 | 1/1 | 5/8 | 13/31
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 4/4 | 4/4 | 4/4 | 6/6 | 1/1 | 8/8 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06664178 0.15 mg/kg (N=2) | PF-06664178 0.30 mg/kg (N=2) | PF-06664178 0.60 mg/kg (N=4) | PF-06664178 1.20 mg/kg (N=4) | PF-06664178 2.40 mg/kg (N=4) | PF-06664178 3.60 mg/kg (N=6) | PF-06664178 4.20 mg/kg (N=1) | PF-06664178 4.80 mg/kg (N=8) | Total (N=31)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06664178 0.15 mg/kg (N=2) | PF-06664178 0.30 mg/kg (N=2) | PF-06664178 0.60 mg/kg (N=4) | PF-06664178 1.20 mg/kg (N=4) | PF-06664178 2.40 mg/kg (N=4) | PF-06664178 3.60 mg/kg (N=6) | PF-06664178 4.20 mg/kg (N=1) | PF-06664178 4.80 mg/kg (N=8) | Total (N=31)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 5 | 8
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 2 | 1 | 0 | 5 | 11
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2 | 2 | 0 | 0 | 6
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Lip blister (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2 | 3 | 0 | 3 | 10
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Palatal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 5
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 5
Chills (General disorders) | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 4 | 9
Early satiety (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Face oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 3 | 1 | 1 | 4 | 0 | 4 | 13
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Local swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 5
Oedema peripheral (General disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 5
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 5
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 4
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 2 | 8
Body temperature increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 4 | 8
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0 | 1 | 1 | 0 | 1 | 7
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 4
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 2 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 3
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Scrotal erythema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 5
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 5
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 4
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 4
Facial wasting (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 6
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 4 | 8
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 5
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3
Red man syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin striae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3

LIMITATIONS AND CAVEATS:
The study was terminated prematurely for business reasons

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.